CLINICAL TRIAL: NCT06508294
Title: Investigation of 8-Week Artificial Intelligence Based Structured Exercise Program in Healthy Adults
Brief Title: 8-Week Artificial Intelligence Based Structured Exercises
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Collaborators: Gulhane Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Tezel Yıldırım Şahan, Associate Professor, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024-180
Record Dates: First submitted 2024-05-15; First posted 2024-07-18 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Health Behavior
Keywords: posture; exercise; artificial intelligence; craniovertebral angle
MeSH Terms: conditions — Health Behavior; Motor Activity

STUDY DESIGN:
Intervention Model Description: 8 week artifical intelligence based posture exercises
Who Masked: Participant
Masking Description: a random list was taken from randomised.org
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 8 week artifical intelligence based posture exercises (Experimental): An artificial intelligence application called "Musclewiki" will be used for healthy adults to continue their exercise training at home. For 8 weeks, exercise will be practiced 3 times a week in the company of a physiotherapist, accompanied by a physiotherapist through artificial intelligence.
  Interventions: Behavioral: 8 week artificial intelligence based posture exercises
- Control (No Intervention): This group of healthy adults will be evaluated before and after 8 weeks and no exercise will be performed.

INTERVENTIONS:
Behavioral: 8 week artificial intelligence based posture exercises — 8 week artificial intelligence based posture exercises
  Arms: 8 week artifical intelligence based posture exercises

SUMMARY:
Posture is defined as the arrangement or orientation of body parts in relation to each other.In this study, it was aimed to examine the effect of an 8-week artificial intelligence-based structured exercise program in healthy adults. It performs measurements on frontal and lateral images of the individual in normal posture Photo of a participant showing how the Posture Screen Mobile app evaluates the horizontal tilt and inclination of the head, shoulders and hips from a frontal view.The craniovertebral angle (CVA) is a measurement of upper cervical posture obtained by calculating the angle between the ear tragus and a horizontal line passing through the spinous process of C7). KVA will be done with Posture Screen Mobile Phone application.Thoracic kyphosis is the anteroposterior curve of the thoracic spine in the sagittal plane and is defined using the Cobb angle.Thoracic kyphosis is the hunching of the spine in the upper back into an extreme external curve due to deformity.An artificial intelligence application called "Musclewiki" will be used for healthy adults to continue their exercise training at home. For 8 weeks, exercise will be practiced 3 times a week in the company of a physiotherapist, accompanied by a physiotherapist through artificial intelligence.

DETAILED DESCRIPTION:
Posture is defined as the arrangement or orientation of body parts in relation to each other. This alignment depends on the effect of gravity, muscle tension and the integrity of the bony structures. Posture disorders, which are now common among healthy young adults, are caused by a number of factors that have emerged in combination with the effects of modern lifestyle.In this study, it was aimed to examine the effect of an 8-week artificial intelligence-based structured exercise program in healthy adults. It performs measurements on frontal and lateral images of the individual in normal posture Photo of a participant showing how the Posture Screen Mobile app evaluates the horizontal tilt and inclination of the head, shoulders and hips from a frontal view.The craniovertebral angle (CVA) is a measurement of upper cervical posture obtained by calculating the angle between the ear tragus and a horizontal line passing through the spinous process of C7). KVA will be done with Posture Screen Mobile Phone application.Thoracic kyphosis is the anteroposterior curve of the thoracic spine in the sagittal plane and is defined using the Cobb angle.Thoracic kyphosis is the hunching of the spine in the upper back into an extreme external curve due to deformity.Lumbar lordosis is the natural inward curve of the spine in the lumbar region. It is an important anatomical feature that maintains the height of the discs in front of the lumbar vertebrae and ensures the stability of the spine.An artificial intelligence application called "Musclewiki" will be used for healthy adults to continue their exercise training at home. For 8 weeks, exercise will be practiced 3 times a week in the company of a physiotherapist, accompanied by a physiotherapist through artificial intelligence.

ELIGIBILITY:
Inclusion Criteria:

* having a smartphone
* volunteering to participate in the study

Exclusion Criteria:

* having a neurological, orthopedic or rheumatologic problem in the spine that will affect its mechanics
* a history of cancer affecting the spine
* a history of any trauma to the spine in the last 6 months
* having vision or hearing problems that may affect the use of artificial intelligence

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
craniovertebral angle measurement | before- after 8 week
  angle degree measurement with telephone application

SECONDARY OUTCOMES:
thoracal kyphosis angle | before-after 8 week
  angle degree measurement with telephone application
lumbal lordosis angle | before-after 8 week
  lumbal lordosis angle degree measurement with telephone application

CONTACTS AND LOCATIONS:
Overall Officials: Tezel Y Şahan, phD, Study Chair — University of Health science
Locations (1):
- University of Health Science, Ankara, Kecioren, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Salsali M, Sheikhhoseini R, Sayyadi P, Hides JA, Dadfar M, Piri H. Association between physical activity and body posture: a systematic review and meta-analysis. BMC Public Health. 2023 Aug 30;23(1):1670. doi: 10.1186/s12889-023-16617-4. PMID 37649076
- [Background] Moustafa IM, Diab AA. The effect of adding forward head posture corrective exercises in the management of lumbosacral radiculopathy: a randomized controlled study. J Manipulative Physiol Ther. 2015 Mar-Apr;38(3):167-78. doi: 10.1016/j.jmpt.2014.11.009. Epub 2015 Feb 20. PMID 25704221
- [Background] Jung SH, Hwang UJ, Kim JH, Gwak GT, Kwon OY. Effect of improved thoracic kyphosis on forward shoulder posture after mobilization in individuals with thoracic hyperkyphosis. Clin Biomech (Bristol). 2022 Jul;97:105707. doi: 10.1016/j.clinbiomech.2022.105707. Epub 2022 Jun 18. PMID 35763888
- [Background] Bruyneel AV, Duclos NC. Effects of the use of mobile phone on postural and locomotor tasks: a scoping review. Gait Posture. 2020 Oct;82:233-241. doi: 10.1016/j.gaitpost.2020.09.014. Epub 2020 Sep 16. PMID 32979702
- [Background] Sepehri S, Sheikhhoseini R, Piri H, Sayyadi P. The effect of various therapeutic exercises on forward head posture, rounded shoulder, and hyperkyphosis among people with upper crossed syndrome: a systematic review and meta-analysis. BMC Musculoskelet Disord. 2024 Feb 1;25(1):105. doi: 10.1186/s12891-024-07224-4. PMID 38302926